CLINICAL TRIAL: NCT02696499
Title: Treatment of Uremic Pruritus With Inhaled PA101B in Patients With End-Stage Renal Disease Requiring Hemodialysis
Brief Title: Treatment of Uremic Pruritus With PA101B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patara Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA101B-UP-02
Record Dates: First submitted 2016-02-25; First posted 2016-03-02 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Uremic Pruritus
Keywords: Uremic pruritus; Pruritus; Chronic itch; Itch; Hemodialysis; End-stage renal disease
MeSH Terms: conditions — Pruritus; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PA101B (Experimental)
  Interventions: Drug: PA101B
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PA101B — 40 mg PA101B administered via inhalation twice daily for 7 weeks
  Arms: PA101B
Drug: Placebo — Matching placebo administered via inhalation twice daily for 7 weeks
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled, parallel-arm, multi-center, Phase 2, proof-of-concept efficacy and safety study in patients with end-stage renal disease requiring hemodialysis.

The purpose of the study is to determine the efficacy and safety profile of PA101B delivered via eFlow high efficiency nebulizer in patients with uremic pruritus who are symptomatic despite using standard treatments.

DETAILED DESCRIPTION:
The symptom score for determining eligibility will be established during the Screening Period (up to 4 weeks) and eligible patients will be randomly allocated in a 2:1 ratio between the active and placebo arms at the baseline visit (Week 0). During the Treatment Period, clinic visits will occur at the end of Weeks 1, 3, 5 and 7. Following completion of the Treatment Period, patients will enter a 2-week Washout Period in both treatment arms.

Routine hemodialysis treatment will continue according to the dialysis unit's standard practice in all patients.

Patients will be allowed to continue to use the same daily doses of pre-randomization H1 antihistamines as well as the same daily doses of any other allowed medications throughout the study.

Blood samples will be collected for various biomarkers. In a subset of patients, additional blood samples will be collected for pharmacokinetic assessments. Clinical safety assessments will be performed at each clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of end-stage renal disease (ESRD) requiring hemodialysis for at least 3 months prior to the Screening Period
* Receiving conventional hemodialysis (i.e., not hemofiltration or hemodiafiltration)
* Pruritus present for at least 6 weeks of Screening
* Mean pruritus severity score on a numerical rating scale (NRS) > 4
* Patient-Assessed Disease Severity Scale Type B or C at Screening
* Documentation of a urea reduction ratio (URR) >65% or single-pooled Kt/V> 1.4 during Screening
* Willing and able to provide written informed consent

Exclusion Criteria:

* Current or recent history of clinically significant medical condition, laboratory abnormality, or illness that could put the patient at risk or compromise the quality of the study data as determined by the investigator
* Myocardial infarction within 6 months or unstable angina, acute coronary syndrome, or interventional coronary procedure within 2 months of Screening
* Upper or lower respiratory tract infection (including sinus infection) within 4 weeks of Screening
* Severely symptomatic cardiopulmonary disease defined by the use of home oxygen treatment, dyspnea at rest or with minimal exertion, uncontrolled arrhythmias (e.g. atrial fibrillation with inadequate rate control), or history of life-threatening arrhythmias (e.g. cardiac arrest or syncope related to arrhythmia)
* Acute exacerbation of asthma or chronic obstructive pulmonary disease resulting in hospitalization or visit to an emergency department or urgent care clinic within 6 months of Screening
* Hospitalization for any medical reason other than for a pre-planned procedure or dialysis access related procedure within the 2 weeks of Screening
* Malignancy requiring active treatment with a systemic drug
* Participation in any other investigation drug study within 4 weeks of Screening
* Current or anticipated use of baclofen, gabapentin, pregabalin and nalbuphine for the treatment of pruritus
* Current or anticipated use of glucocorticoids administered intravenously, orally, or transdermally
* Pregnant or breastfeeding females, or if of child-bearing potential unwilling to practice acceptable means of birth control or abstinence during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Itching intensity | 7 weeks
  Numerical rating scale (NRS)

SECONDARY OUTCOMES:
Pruritus-specific quality of life (QoL) | 7 weeks
  Skindex-10
Pruritus-specific sleep quality | 7 weeks
  Itch MOS
Assessment of depression | 7 weeks
  Beck Depression Inventory-II
Patient Global Impression of Change (PGIC) | 7 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Arizona Kidney Disease and Hypertension Center, Phoenix, Arizona
  - US Renal Care, Pine Bluff, Arkansas
  - Valley Renal Medical Group, Northridge, California
  - North America Research Institute, San Dimas, California
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Boise Kidney and Hypertension Institute, Meridian, Idaho
  - Fresenius Medical Care of Evergreen Park, Evergreen Park, Illinois
  - Renal Medicine Associates, Albuquerque, New Mexico
  - US Renal Care, Gallup, New Mexico
  - Ridgewood Dialysis Center, Ridgewood, New York
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264